CLINICAL TRIAL: NCT06361914
Title: Digital CBT-I for Patients With Chronic Pain and Insomnia (The Back2Sleep Trial). A Randomized Controlled Trial
Brief Title: Digital CBT-I for Patients With Chronic Pain and Insomnia
Acronym: Back2Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); University of Southern Denmark (Other); University of Aarhus (Other); Odense Patient Data Explorative Network (Other); T&W Engineering A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2314393
Record Dates: First submitted 2024-03-27; First posted 2024-04-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Insomnia
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Sleep hygiene education (Active Comparator): Sleep hygiene education is the commonly delivered treatment for insomnia in patients with chronic pain. The digital sleep hygiene education treatment in the Hvil® app includes the sleep hygiene education element that entails specific information relating to lifestyle (diet, exercise, substance use) and environmental factors (light, noise, temperature) that may interfere with or promote sound sleep. Sleep hygiene education also includes specific sleep facilitating recommendations, such as avoiding visual access to a clock in the bedroom, regular sleep scheduling, avoiding long daytime naps, and limiting alcohol, caffeine, and nicotine intake. Parallel to engaging with this element, participants are asked to fill in a sleep diary during the intervention's entire course.
  Interventions: Behavioral: Digital Sleep hygiene education
- Digital CBT-I (Experimental): The digital CBT-I intervention in the Hvil® app is designed to be completed over a period of nine weeks (5 weeks with the components described below and 4 weeks with maintenance of new habits), and is based on the current consensus concerning non-pharmacological treatment of insomnia including five treatment components (sleep restriction, stimulus control, deactivation/relaxation training, cognitive therapy, sleep hygiene education). Each treatment component consists of an information module (i.e., content and purpose of the specific component), assessment module (i.e., assessment of the severity of the "problem" addressed by the component), application module (i.e., specific information on different types of exercises the participant should engage in), and evaluation module (i.e., assessment of the treatment gain). Participants are encouraged to complete the information and assessment module in one streak, estimated to last 30-60 minutes.
  Interventions: Behavioral: Digital CBT-I

INTERVENTIONS:
Behavioral: Digital CBT-I — Sleep restriction includes behavioral instructions to limit the time spent in bed to increase sleep drive and further reduce time awake in bed.
  Stimulus control therapy entails behavioral instructions to strengthen the association between bed and sleep and to eliminate conditioning of non-sleep behavior and bed.
  Deactivation/relaxation training involves methods to reduce somatic tension and limit intrusive thought processes that interfere with sleep.
  Cognitive therapy helps to identify, challenge, and modify dysfunctional beliefs about sleep.
  Sleep hygiene education entails specific information relating to lifestyle and environmental factors that may interfere with or promote sound sleep. Sleep hygiene education also includes specific sleep facilitating recommendations, such as avoiding visual access to a clock in the bedroom, regular sleep scheduling, avoiding long daytime naps, and limiting alcohol, caffeine, and nicotine intake.
  Arms: Digital CBT-I
Behavioral: Digital Sleep hygiene education — Sleep hygiene education entails specific information relating to lifestyle (diet, exercise, substance use) and environmental factors (light, noise, temperature) that may interfere with or promote sound sleep. Sleep hygiene education also includes specific sleep facilitating recommendations, such as avoiding visual access to a clock in the bedroom, regular sleep scheduling, avoiding long daytime naps, and limiting alcohol, caffeine, and nicotine intake.
  Arms: Digital Sleep hygiene education

SUMMARY:
Chronic pain constitutes an increasing health and social burden. More than 50% of patients with chronic pain report insomnia, and patients with comorbid insomnia often report stronger and widespread pain, compared to those who are sleeping well. Sleep disturbances are often considered a consequence to chronic pain. This means that insomnia is often overlooked or ineffectively managed with hypnotics or advice on sleep hygiene. Therefore, efficacious, easily accessible, and safe alternatives to the current pharmacological treatments for patients with chronic pain and insomnia are needed. Cognitive behavioral therapy for insomnia (CBT-I) is a cost-effective and safe treatment for insomnia and is recommended as first-line treatment. While highly efficacious, the challenge is to deliver CBT-I to those in need. The main barriers of face-to-face delivered CBT-I are availability of trained therapists, costs, as well as physical and geographical constraints.

The primary aim of this randomized controlled clinical superiority trial is to investigate whether digitally-delivered CBT-I has a greater effect on insomnia and pain than digitally-delivered sleep hygiene education in patients with chronic pain and comorbid insomnia.

Secondary objectives are to a) explore whether the pain-relieving effect is mediated by a change in physiological markers of sleep quality, b) whether health care cost and use of medications at 12 months are reduced after digital CBT-I, and c) to explore the effectiveness of digital CBT-I compared with sleep hygiene education on:

1. Physiological sleep metrics (recorded with ear EEG in subsample of 60 patients).
2. Self-reported sleep quality.
3. Quality of life.
4. Physical and mental health.
5. Thoughts and beliefs about sleep and pain.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of digital CBT-I for improving sleep (i.e. reducing insomnia severity) and reducing pain intensity in patients with chronic pain and comorbid insomnia. To achieve this goal, the investigators will perform a randomized controlled single-blind clinical superiority trial. Participants will be randomized with an allocation 1:1 ratio into a digital CBT-I group and a sleep hygiene education group. Both groups will use the Hvil® app, but the amount of content will be different. Using a data manager not affiliated with the project through the Open Patients data Exploratory Network (OPEN) at Odense University Hospital, the randomization will be implemented in the program REDCap. The data manager will prepare the randomization list in REDCap. The computer algorithm will use permuted-block randomization of 2, 4 and 6 individuals. No stratifications will be applied to the randomization.

After inclusion, participants will receive an unique randomization key to impute in the Hvil® app according to the abovementioned procedure to receive either digital CBT-I or sleep hygiene education for 9 weeks. This Hvil® App platform is used for both treatments to ensure that only the contents is different, but the form of delivery is the same. All patient reported data will be filled in directly to the eCRF via an online questionnaire using REDCap. Statistical analyses will be blinded to treatment allocation.

Sample size estimation:

Minimal clinical important difference for insomnia severity is 5 point. With an estimated SD for change of 2 times the minimal clinical important difference (SD=10) for patients with chronic pain and insomnia, power of 80%, an alpha value of 0.05, a minimum of 63 participants in each group is required.

Minimal clinical important difference for pain intensity is 15% corresponding to a change of 1.0 points in this population. With a SD for change of 2.0 for patients with chronic pain and insomnia, power of 80%, an alpha value of 0.05, a minimum of 63 participants in each group is required.

With an expected drop-out of 30% the investigators plan to recruit 160 participants (80 for each group).

Stopping rules: This trial has two stopping rules. Inclusion will stop December 31st 2025. In the event that 130 patients have completed the 9 weeks follow-up before 160 patients have been recruited the investigators will stop recruitment of further participants.

All participants that are withdrawn from the study will be encouraged to complete all visits as scheduled. Participants that are withdrawn from the treatment will not be replaced and will be included in the intention-to-treat population. According to the sample size calculation, the investigators will include participants enough to tolerate a drop-out rate of up to 30%. Both intention-to-treat and per protocol analysis will be performed and compared to assess the robustness of the primary analysis.

Statistical methods:

Difference in change from baseline to 9 weeks in the two primary outcomes (ISI score or mean NRS pain in last 7 days, both being continuous variables) between the digital CBT-I group and the sleep hygiene education group will be estimated using a mixed linear model approach with ISI and NRS pain as outcomes, time, treatment arm (digital CBT-I or sleep hygiene education), and the interaction between time and treatment arm as fixed effects. Both participant specific intercept and slope will be considered as random effects. The model will be adjusted for ISI score or NRS pain at baseline, respectively. The error variance will be allowed to vary over time and across the two arms. Interactions will be parametrized as time dependent treatment effects such that the treatment effect at week 9 corresponds directly with the efficacy parameter of interest. The treatment effect will be expressed as the gain in reduction observed in the digital CBT-I arm, i.e. a positive number expresses a favoring of the intervention. The pre-specified effectiveness analyses will be based on the intention-to-treat (ITT) principle, which includes all participants that are assessed and randomized at baseline. In the case of missing data during the 9-week trial, repeated measures linear mixed models will take this into account automatically, under the assumption that data is missing at random.

For the statistical assessment of the two primary outcomes (ISI and pain intensity), the investigators will apply a sequential test procedure to compare the effect of the two treatments (CBT-I vs. sleep hygiene education) on ISI severity in the first step and the effect on pain intensity in the second step. This means that statistical significance in the second step will only be assessed if statistical significance has been reached in the first step . The investigators use this approach as it seems unlikely that these interventions has direct effect on pain, but rather work through improved sleep. The significance level is set to 5%.

In responder analysis, a responder is defined as a patient who report a more than 30% and 50% decrease in insomnia or pain after 9 weeks. Proportion of responders between treatment groups will be expressed by adjusted odds ratios. These will be based on a logistic regression model with treatment, baseline value of pain intensity and insomnia severity, and sex as covariates.

A detailed statistical analysis plan (SAP) will be made publicly available before the statistical analysis is initiated.

ELIGIBILITY:
Inclusion Criteria:

For a participant to be eligible, all inclusion criteria must be answered "yes":

* Age ≥ 18 years.
* Understand and write Danish.
* Have smartphone access.
* Pain for 3 months or longer.
* Pain must be present on 'most days' or 'every day' within the past 3 months (will be checked by the question: 'In the past 3 months, how often did you have pain? - response options: 'never'; 'some days'; 'most days'; 'every day').
* Pain must limit life or work activities on 'some days', 'most days', or 'every day' within the past 3 months (will be checked by the question: 'In the past 3 months, how often did your pain limit your life or work activities - response options: never, some days, most days, every day
* Average pain intensity equal to or higher than 4 on a 0-10 Numeric Rating Scale [NRS] in the past 7 days (ranging from 'no pain' to 'worst imaginable pain').

Insomnia symptoms (Insomnia Severity Index (ISI) score > 10; moderate insomnia).

Exclusion Criteria:

For a participant to be eligible, all exclusion criteria must be answered "no":

* Pregnancy or lactation (Pregnancy is screened for through self-reporting as no risks regarding pregnancy have been identified for the described study procedures).
* Does not have daily assess to smartphone/tablet
* Night shift during the time of the CBT-I treatment.
* Currently receiving pharmacological treatment for insomnia (e.g. benzodiazepines, hypnotics etc.).
* Severe psychiatric/somatic illnesses of relevance of their sleep (reported by participant).
* Diagnosed sleep disorders (e.g., OSA, narcolepsy).
* Does not have E-boks.
* Known abuse of alcohol or other substances.
* Suicide and self-harm thoughts (reported by participant).
* People judged incapable, by the investigator, of understanding the participant instruction or who are not capable of carrying through the investigation.

For the EEG subgroup only (60 patients):

* Age ≥ 65 years
* Anatomy of the outer ear making it impossible to do ear EEG monitoring.
* Ear piercings that are not compatible with ear EEG.
* Previous stroke or cerebral haemorrhage and any other structural cerebral disease.
* Teeth grinding (bruxism).
* Allergic contact dermatitis caused by metals or generally prone to skin irritation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | Difference in change between groups from baseline to 9 weeks.
  Insomnia will be assessed with the Insomnia Severity Index (ISI), which is a brief 7 item patient-reported instrument with a score ranging from 0-28 (0=best;28=worst)
Average pain intensity during the last 7 days | Difference in change between groups from baseline to 9 weeks
  Average pain intensity during last 7 days will be assessed on a 0-10 Numeric Rating Scale (NRS) (ranging from 'no pain to 'worst imaginable pain')

SECONDARY OUTCOMES:
The trajectory of ISI severity scores | Baseline, after 4 weeks, after 9 weeks
  The trajectory of ISI scores from baseline, at 4 weeks and 9 weeks
30% ISI responders | Change from baseline to 9 weeks
  Difference in number of patients with more than 30% improvement in ISI severity score from baseline to 9 weeks
50% ISI responders | Change from baseline to 9 weeks
  Difference in number of patients with more than 50% improvement in ISI severity score from baseline to 9 weeks
Weekly pain intensity score trajectory | Weekly from baseline to 9 weeks
  The trajectory of weekly NRS pain intensity scores from baseline to 9 weeks
30% pain intensity responders | Change from baseline to 9 weeks
  Difference in number of patients with more than 30% improvement in pain intensity from baseline to 9 weeks
50% pain intensity responders | Change from baseline to 9 weeks
  Difference in number of patients with more than 50% improvement in pain intensity from baseline to 9 weeks
Global Perceived Effect (GPE) for sleep | After 9 weeks
  Assessment of overall change in insomnia from baseline to 9 weeks. Participants will be asked at 9 weeks: 'How is your insomnia now compared to when you entered this study', with 5 response options (much worse, worse, almost the same/unchanged, improved, much improved)
Global Perceived Effect (GPE) for pain | After 9 weeks
  Assessment of overall change in pain from baseline to 9 weeks. Participants will be asked at 9 weeks: 'How is your pain now compared to when you entered this study', with 5 response options (much worse, worse, almost the same/unchanged, improved, much improved)
Sleep Quality | Baseline, after 4 weeks and after 9 weeks
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI), which is developed to provide a reliable, valid and standardized measure of sleep quality. The PSQI consists of 19 items with 15 multiple choice questions and 4 open-ended questions. The 19 items form the basis a global score. The seven components evaluated by the PSQI are: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications and daytime dysfunction. Each component has a score ranging from 0 to 3 yielding a total score of 21, with higher scores reflecting worse sleep difficulties
Physical and Mental Health | Baseline and after 9 weeks
  Physical and Mental Health will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS-10) Global Health questionnaire version 1.2. Difference in change in physical and mental health scores between treatment groups from baseline to 9 weeks. PROMIS-10 consist of 10 questions concerning different aspects of global health. The first 9 questions are score on a Likert scale with 5 response options, and the last question asks about pain using a 0-10 numeric rating scale
Sleep diary | Daily for 7 nights at baseline and after 9 weeks
  Sleep diary (total sleep time and sleep efficiency) implemented in the Hvil® app.
Thoughts about sleep and pain | Baseline, after 4 weeks and after 9 weeks
  Thoughts about sleep and pain via the Pain-Related Beliefs and Attitudes about Sleep (PBAS) questionnaire. PBAS consist of 10 items.
Thoughts about sleep | Baseline, after 4 weeks and after 9 weeks
  Thoughts about sleep via the Dysfunctional Beliefs and Attitudes About Sleep (DBAS) Questionnaire. DBAS consist of 16 questions.
Treatment compliance | After 9 weeks
  To explore compliance with the treatment arms the interaction with the Hvil App will be explored. This will be reported in terms of time/frequency of using with the app over the 9 weeks.
Health-related quality of life - mobility | Baseline and after 9 weeks
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) mobility domain; asking the participants to rate their mobility on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems
Health-related quality of life - self care | Baseline and after 9 weeks
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) self care domain; asking the participants to rate their ability for self care on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - usual activities | Baseline and after 9 weeks
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) usual activities domain; asking the participants to rate their ability to perform usual activities on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - pain/discomfort | Baseline and after 9 weeks
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) pain/discomfort domain; asking the participants to rate their level of pain or discomfort on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - anxiety/depression | Baseline and after 9 weeks
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) anxiety/depression domain; asking the participants to rate their level of anxiety or depression on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - global | Baseline and after 9 weeks
  Measured by European Quality of Life Visual Analogue Scale (EQ-VAS), which asks the participant to rate their overall health 'today' on a 0-100 VAS. A higher score indicates a better quality of life.

OTHER OUTCOMES:
Age | Baseline
  The age of the participant will be calculated using the date of randomisation and the date of birth.
Sex | Baseline
  The sex of the participant assigned at birth (male or female)
Chronic pain | Baseline
  Chronic pain will be assessed using the Graded Chronic Pain Scale Revised (GCPS-R) questionnaire. The GCPS-R is a brief, freely available questionnaire that assesses frequency and severity of pain and its impact. The GCPS-R uses 5 items to categorize pain into no chronic pain, mild chronic pain, bothersome chronic pain, and high-impact chronic pain
Ethnicity | Baseline
  The categories for data on ethnicity are White, Asian, Black or African American, other
Height | Baseline
  Self-reported in centimeter
Weight | Baseline
  Self-reported in kilograms
Marital status | Baseline
  Self-reported marital status
Level of education | Baseline
  The categories for level of education are compulsory education, upper secondary, bachelor degree, master degree, Phd degree
Pain distribution | Baseline
  Using a pain drawing, patients will be classified into different pain groups at baseline: widespread pain, referred/radiating back pain patterns, regional and localized pain.
Medical history and concomitant illnesses | Baseline
  Self-reported medical history and concomitant illnesses relevant to the investigation will be recorded in the eCRF by a trained study nurse during the information visit. A clinically significant worsening of a concomitant illness will be reported as an AE
Concomitant medication | Baseline
  Self-reported concomitant medication will be recorded in the eCRF by a trained nurse during the information visit.
Health-related quality of life - mobility | After 12 months
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) mobility domain; asking the participants to rate their mobility on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - self care | After 12 months
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) self care domain; asking the participants to rate their ability for self care on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - usual activities | After 12 months
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) usual activities domain; asking the participants to rate their ability to perform usual activities on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - pain/discomfort | After 12 months
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) pain/discomfort domain; asking the participants to rate their level of pain or discomfort on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - anxiety/depression | After 12 months
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) anxiety/depression domain; asking the participants to rate their level of anxiety or depression on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems.
Health-related quality of life - global | After 12 months
  Measured by European Quality of Life Visual Analogue Scale (EQ-VAS), which asks the participant to rate their overall health 'today' on a 0-100 VAS. A higher score indicates a better quality of life.
Insomnia Severity | After 6 months
  Insomnia will be assessed with the Insomnia Severity Index (ISI), which is a brief 7 item patient-reported instrument with a score ranging from 0-28 (0=best;28=worst)
Average pain intensity during the last 7 days | After 6 months
  Average pain intensity during last 7 days will be assessed on a 0-10 Numeric Rating Scale (NRS) (ranging from 'no pain to 'worst imaginable pain')
Medication use | After 12 months
  Proportion of participants using analgesics and sleep medication will be explored using data from the prescription database.
Economical evaluation | after 12 months
  The healthcare costs will be obtained from linking the trial data to Danish health registries. The healthcare costs of treatment will be reported in euro.
Time from sleep onset until final awakening (TST) from Ear EEG in subgroup of 60 patients | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Sleep efficiency (SE) from Ear EEG in subgroup of 60 patients | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM). SE is the ratio of TST to time in bed / 100%
Sleep onset latency (SOL) from Ear EEG in subgroup of 60 patients | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Wake after sleep onset (WASO) from Ear EEG in subgroup of 60 patients | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
REM sleep latency from Ear EEG in subgroup of 60 patients | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Time from sleep onset until first epoch of REM stage sleep from Ear EEG | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Amount of wake and stage N1, N2, N3, and R sleep as a percentage of SPT from Ear EEG | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Number of awakenings within TST from Ear EEG | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Arousal index which is number of arousals per hour from Ear EEG | Difference in change in sleep metric between treatment groups from baseline to 8 weeks.
  Difference in change in sleep metric between treatment groups (digital CBT-I [n=30] vs.sleep hygiene education [n=30]) from baseline to 8 weeks. Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Ease-of-use and Comfort with ear EEG | 5 nights at baseline and 5 nights at week 8
  Three 0-10 questions are used: 1) How did you experience falling asleep with the ear EEG device, 2) How did you experience sleeping with the ear EEG device?, 3) How would you rate your experience of soreness or discomfort in your ears after sleeping with the device? A lower sum score is worse.
Ear EEG adverse device effects | Baseline and 8 weeks
  Any adverse device effect defined as an adverse effect related to the use of the ear EEG

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Vægter, PhD, Principal Investigator — University Hospital Odense
Locations (1):
- Pain Center, Department of Anesthesiology and Intensive Care Medicine, University Hospital Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsen MLS, Thorlund JB, Zachariae R, Vach W, Bendix L, Jespersen J, Kidmose P, Parsons C, Kidholm K, Vaegter HB. Digitally delivered cognitive behavioral therapy for insomnia (CBT-I) for patients with chronic pain and insomnia (The Back2Sleep Trial): study protocol for a randomized controlled trial. Trials. 2025 Aug 15;26(1):292. doi: 10.1186/s13063-025-09013-3. PMID 40817235